CLINICAL TRIAL: NCT02605603
Title: Effect of Two Different Therapeutic Interventions: SRT in Comparison to ERT on Immune Aspects and Bone Involvement in Gaucher Disease
Brief Title: SRT in Comparison to ERT on Immune Aspects and Bone Involvement in Gaucher Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 15-LDRTC-02
Record Dates: First submitted 2015-09-09; First posted 2015-11-16 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Gaucher Disease
Keywords: Gaucher Type 1, Gaucher Type 2, Gaucher Type 3
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project is expected to elucidate role of different therapeutic interventions: SRT in comparison to ERT in influencing immune aspects of GD pathology, as well as bone involvement.

DETAILED DESCRIPTION:
Introduction

Lysosomes are small, cytoplasmic organelles that contain several acid hydrolase enzymes. These enzymes break down foreign materials and cellular debris allowing the lysosomes to act as recycling centers for the cells. Following DNA transcription, lysosomal enzymes are produced in the endoplasmic reticulum and targeted to lysosomes by specific recognition markers. If one of the enzymes is absent or if its function is diminished due to either an altered amino acid sequence of the protein or defective intracellular trafficking, the macromolecules metabolized by the specific enzyme will gradually accumulate in the lysosomes. Abnormal substrate storage leads to cellular dysfunction followed by cell death ultimately manifesting as tissue damage and organ failure.

Gaucher disease (GD) is a lysosomal storage disorder caused by a genetic deficiency of the lysosomal enzyme glucocerebrosidase. GD leads to accumulation of glycosphingolipids in various tissue systems, most notably in cells of mononuclear phagocyte system resulting in a wide range of heterogenous phenotypic effects in the affected individuals. Clinical manifestations of GD affect across multiple organs ranging from immune dysregulations, splenomegaly to bone crises and osteoporosis. Carrier frequency is 1 in 200 for the general population with an incidence of 1 in 60,000. However, in certain populations, such as Ashkenazi Jews, the incidence could be as high as 1 in 1,000.

Background and Significance

Macrophage directed Enzyme replacement therapy (ERT) has been the most accepted form of treatment for GD. However there are still unmet needs in treating all aspects of GD using ERT. As an alternative to ERT, substrate reduction therapy (SRT) was developed using glucosylceramide synthase inhibitors. While ERT is devised to target macrophages which are the most affected cell types, SRT is meant to reach broad cell types. It is vital to know how each form of therapy acts on different cell types and tissues while choosing to administer either form of treatment on individual patients. Our preliminary immune phenotyping results reveal that patients with GD undergoing treatment manifest various kinds of persistent immune dysregulations. Information regarding which type of therapy works better in controlling these dysregulations would give valuable information in treatment options. In-depth analysis on peripheral blood would shed light as to how various components of immune system are being affected with either form of treatment.

The investigators will address this issue from two aspects: a) Evaluate cytokine profile from plasma to see if the reported pain correlates with a particular cytokine profile. b) Assess if the extent of bone disease could be predicted or explained using markers from peripheral blood in relation to pathways involved in bone remodeling. The findings from individual GD patients would be compared in parallel to their disease severity and bone density findings.

In this study, the effects of ERT vs SRT will be closely monitored and compared, particularly keeping in mind immunological aspects as well as bone remodeling. For this, in-depth immunophenotyping of patients being administered these forms of therapy to evaluate various immune cell types including T-, B- and NK cell, monocyte and dendritic cell fractions from peripheral blood using multi-parametric flow cytometry will be performed. In addition to these the investigators will like to assess the macrophage activation using assays for secreted CCL18 and chitotriosidase as well as study the cytokine profile from plasma to evaluate their contribution to bone pain/crisis. In order to investigate if the extent of bone remodeling could be predicted or explained using markers from peripheral blood, expression of RANK/RANKL pathway components would be assessed on relevant immune cell types. Cell based in vitro assays would be developed and utilized to study differentiation and macrophage function. The results from individual GD patients would be compared in parallel to their disease severity and bone density findings. This proposal is highly significant and innovative, because this study is expected to provide insights into how each form of therapy influences the immune dysregulations, macrophage function and their effects on bone crisis in Gaucher patients undergoing ERT vs SRT. Insight regarding which type of therapy works better in controlling these dysregulations would give valuable information in treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Gaucher disease
2. Subjects on SRT using Cerdelga ( must fulfil the pharmacogenomics criteria for Cerdelga)

Exclusion Criteria:

1. Unconfirmed diagnosis of Gaucher disease
2. Subject or guardian unable to provide consent
3. Any chronic immunosuppressive state or therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Gaucher disease, and are currently on Enzyme replacement therapy (ERT) or on Substrate reduction therapy (SRT).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Delineate T-, B- and NK cell fractions as well as dendritic cell and monocyte numbers and compare between patients undergoing ERT vs. SRT. | 2 Years
  We will utilize multicolour flow cytometry using cell surface markers to perform detailed analysis of various components of immune system. Activation of monocytes/macrophages per se would be measured using secreted cytokines like CCL18 and chitotriosidase from plasma.

SECONDARY OUTCOMES:
Comparative effects on skeletal involvement in individual Gaucher patients correlates with their disease severity and bone involvement. | 2 Years
  Bone mineral deposition will be examined by Alizarin Red staining.

OTHER OUTCOMES:
The effect of Enzyme Replacement Therapy vs. Substrate Replacement Therapy. | 2 years
  Monocytes would be identified as CD45+/CD14+ fraction from peripheral blood in GD patients undergoing ERT or SRT and compared to non- Gaucher controls.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, MD, Principal Investigator — Study Principle Investigator
Locations (1):
- O&O Alpan, LLC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: company information — http://www.ldrtc.org